CLINICAL TRIAL: NCT00186004
Title: Correlation Between Continuous Glucose Monitoring and Intermittent Glucose Monitoring Values and Pregnancy Outcomes
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: Santa Clara Valley Health & Hospital System (Other)
Responsible Party: Yasser Yehia El-Sayed, Stanford University School of Medicine
Other Study IDs: 78694
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2011-06

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Continuous Glucose Monitor — Subjects are fitted with a CGM system and perform self blood glucose measures three or more times per day for 3 days.
  Other Names: Paradigm CGM and FreeStyle Navigator blood glucose monitor.

SUMMARY:
We wish to find out if in non-diabetic pregnancies, as well as diabetic pregnancies, additional data obtained by Continuous Glucose Monitoring improves perinatal risk prediction.

DETAILED DESCRIPTION:
Patients are recruited for 3 day continuous glucose monitoring (CGM) plus self-blood glucose monitoring followed by routine diabetes screening at 26-28 weeks gestation to determine if maternal blood glucose excursions correlate with deviation from optimized birth weight.

ELIGIBILITY:
Inclusion Criteria:

- Pregnant patients under 28 weeks gestation

Exclusion Criteria:

- Pre-gestational diabetes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant patients 18 years or older, less than 28 weeks gestation without pregestational diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2002-12; Primary Completion 2006-09 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Birthweight centile | Delivery

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Yehia El-Sayed, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States